CLINICAL TRIAL: NCT00954733
Title: A Comparison of the Detection of Hypoventilation During Deep Sedation Utilizing Nasal End Title CO@ Versus Transcutaneous CO2 Measurement Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Principal Investigator, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00004382
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-06

CONDITIONS: Surgery; Hypoventilation
Keywords: Hysteroscopic surgery; Hypoventilation; Co2; Transcutaneous Co2 Monitor
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (Experimental): All participants, one arterial blood draw
  Interventions: Other: Arterial blood draw

INTERVENTIONS:
Other: Arterial blood draw — One arterial blood draw

SUMMARY:
The estimation of the partial pressure of carbon dioxide (PCO2) in the arterial blood is used to judge the adequacy of ventilation during spontaneous and controlled ventilation. Although the gold standard for monitoring PCO2 remains arterial blood gas sampling, this requires an invasive procedure and provides only an intermittent estimate of what is frequently a continuously changing value. The solution to this problem has been the development and validation of accurate noninvasive monitoring techniques which provide a continuous intraoperative estimate of PCO2.The most commonly used noninvasive technique to monitor PCO2 is measurement of the end tidal CO2 (PECO2) . However, sampling errors and patient -related issues such as ventilation-perfusion mismatch, patient positioning or decreases in pulmonary blood flow may influence the accuracy of PECO2 monitoring (1-3). Nasal capnography has been proved to be an accurate monitor during the post-operative period (4) but its ability to accurately detect hypoventilation associated with deep sedation has not been studied.

According to the American Society of Anesthesiologist standards for basic monitoring, continuous capnography is required for all patients undergoing general anesthesia but it is optional for MAC/sedation cases. The need for CO2 monitoring has been studied by other medical specialties that use procedural sedation, including gastroenterology (12) and emergency medicine (13, 14) and many specialties now recommend capnography as a standard monitor.

Patients receiving supplemental oxygen may experience significant persistent hypoventilation leading to progressive hypercarbia and acidosis which may go undetected for a significant time interval since the routinely monitored SpO2 may be maintained within normal range. A recent study has shown that despite the fact that end tidal CO2 is reliable in detecting apnea , increasing oxygen flow rates decrease the amplitude of measured CO2, probably via dilution, making the quantitative value less reliable as an assessment of adequacy of ventilation (15). Furthermore, during hypoventilation there is reduced alveolar ventilation and the end tidal CO2 is not a true reflection of arterial CO2.

Transcutaneous measurement of PCO2(PtcCO2) is a non-invasive method of measuring PCO2 that has been used much less frequently due to technical difficulties with earlier transcutaneous electrodes. Preliminary studies of the reliability of the current PtcCO2 electrodes (TOSCA, Linde Medical Sensors, and Basel, Switzerland) have shown good correlation of arterial and transcutaneous measurements in both adult volunteers and anesthetized subjects (5). PtcCO2 is measured with a sensor attached by a low pressure clip to an earlobe. The sensor probe heats the earlobe to 42 degrees Celsius to enhance blood flow. The current sensors have also been evaluated in anesthetized children (7, 8), anesthetized adults (9, 10) and critically ill neonates (11) and all these studies revealed a good correlation between PtCO2 and PaCO2.

DETAILED DESCRIPTION:
A group of _40 patients scheduled to undergo Hysteroscopy surgery with deep sedation will be studied. Standard monitors will be utilized. Additionally a transcutaneous CO2 electrode will be attached to the ear lobe and a BIS monitor will be applied to the forehead.

The anesthetic management will be left to the discretion of the anesthesia provider (Anesthesia resident or CRNA, under the supervision of a faculty attending anesthesiologist).All patients will receive supplemental oxygen at 3L/ minute via nasal cannula, to maintain oxygen saturation greater than 90%.

Both the end tidal CO2 (ETCO2) and transcutaneous CO2 (TcCO2) (Linde Medical Sensors, Basel , Switzerland ) will be calibrated before use, according to the manufacturer's instruction.. The anesthesia provider will be blinded to the TcCO2 monitor but will have access to the ETCO2 values. The ETCO2 and TcCO2 values will be recorded simultaneously by an independent observer.

One arterial blood samples will be collected from each subject for measurement of PaCO2 at a deep level of sedation defined by a modified Ramsey score greater or equal to 5 (1= anxious/agitated/restless; 2= cooperative/oriented/tranquil; 3= drowsy/responds to commands only; 4= brisk response to shaking/loud sound; 5= sluggish response to shaking/loud sound; 6= no response) The ETCO2 and .TcCO2 will be recorded throughout the time of obtaining the blood sample every 15 seconds and the mean value will be used for comparison. Hypoventilation will be defined as a PaCO2 level greater than 45mmHg.

Sedation score (OASS) will be recorded on admission to recovery area. Time to meet discharge criteria will be recorded.

The experimental procedures: ABG draw, ETCO2 monitor placement on the ear, 2 Ramey scale assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years of age
* Sex: Non-pregnant, Female
* ASA PS: I, II
* Surgery: Elective Hysteroscopy surgery
* Consent: Obtained

Exclusion Criteria:

* Age < 18 years old
* Patients who refuses participation
* History of lung disease
* History of Obstructive sleep apnea

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert McCarthy, PharmD, Study Director — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Whitesell R, Asiddao C, Gollman D, Jablonski J. Relationship between arterial and peak expired carbon dioxide pressure during anesthesia and factors influencing the difference. Anesth Analg. 1981 Jul;60(7):508-12. PMID 6787952
- [Background] Yamanaka MK, Sue DY. Comparison of arterial-end-tidal PCO2 difference and dead space/tidal volume ratio in respiratory failure. Chest. 1987 Nov;92(5):832-5. doi: 10.1378/chest.92.5.832. PMID 3117500
- [Background] Grenier B, Verchere E, Mesli A, Dubreuil M, Siao D, Vandendriessche M, Cales J, Maurette P. Capnography monitoring during neurosurgery: reliability in relation to various intraoperative positions. Anesth Analg. 1999 Jan;88(1):43-8. doi: 10.1097/00000539-199901000-00009. PMID 9895064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were approached in the pre operative area sequentially.
Groups:
- All Participants: All participants undergoing surgery
Period: Overall Study
Arm/Group | All Participants
Started | 40
Completed | 39
Not Completed | 1
Not completed — blood gas machine did not work | 1

BASELINE CHARACTERISTICS:
Population: 42 possible participants between 18-65 years of age were approached to participate in the study . 40 gave written informed consent.
Groups:
- All Participants: All participants in the study
Arm/Group | All Participants
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 42 [27 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: TcCo2 vs PACo2 Difference
Description: Evaluate the correlation between PaCO2- TcCO2 in detecting hypoventilation for patients undergoing deep sedation Absolute mean difference between TcCo2 and the PA Co2
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | All Participants
Number analyzed (Participants) | 39
mmHG | 3.2 (2.6)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
We only included healthy, female subjects without significant co-morbidities which limit our ability to generalize our findings to elderly and sicker patients who bay benefit the most from this monitoring.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No